CLINICAL TRIAL: NCT03091816
Title: Dynamic Perfusion Computed Tomography Changes After Stereotactic Body Radiation Therapy for Localized Non-small Cell Lung Cancer
Brief Title: Dynamic Perfusion Computed Tomography in Patients With Localized Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Society of Thoracic Radiology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2N-16-1; NCI-2016-01420 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2N-16-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Stage IA Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Diagnostic (DPCT): Patients undergo DPCT at baseline, during SBRT (after 2 of 3 fractions or 3 of 5 fractions), and then at 1 and 3 months post stereotactic body radiation therapy.
  Interventions: Device: Computed Tomography Perfusion Imaging; Other: Laboratory Biomarker Analysis; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Device: Computed Tomography Perfusion Imaging — Undergo DPCT
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT

SUMMARY:
This pilot clinical trial studies the changes in dynamic perfusion computed tomography images before, during, and after stereotactic body radiation therapy in patients with stage I-II non-small cell lung cancer that has not spread to other parts of the body. Diagnostic imaging procedures, such as dynamic perfusion computed tomography, measure blood flow through tumors. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue. Giving dynamic perfusion computed tomography images before, during, and after stereotactic body radiation therapy may help better understand how radiation therapy works to stop tumor growth in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe perfusion computed tomography (CT) parameters and their changes in non-small cell lung cancer (NSCLC) tumors prior to, during, 1 month after, and 3 months after stereotactic body radiation therapy (SBRT).

SECONDARY OBJECTIVES:

I. To correlate tumor perfusion parameters with clinical tumor response on follow up per standard of care.

TERTIARY OBJECTIVES:

I. To correlate changes in serum levels of deoxyribonucleic acid (DNA) methylation and circulating tumor cell (CTC) with clinical response rates and perfusion parameters.

OUTLINE:

Patients undergo dynamic perfusion computed tomography (DPCT) at baseline, during SBRT (after 2 of 3 fractions or 3 of 5 fractions), and then at 1 and 3 months post stereotactic body radiation therapy.

After completion of study, patients are followed up at 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven non-small cell lung cancer
* Minimum tumor dimension >= 1 cm (preferably >= 2 cm)
* No clinical evidence of nodal disease (N1-N3) as assessed by CT and/or positron emission tomography (PET)/CT
* Zubrod performance status 0-2
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* No prior radiation to the same area
* No concurrent chemotherapy
* Evaluated by radiation oncologist to be appropriate SBRT candidate and scheduled to undergo SBRT as part of their care
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients with tumors < 1 cm
* Patients with nodal disease or distant metastatic disease
* Patients may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not be pregnant
* Patients with allergies to iodinated contrast not amenable to pre-medication
* Patients who are not able to lie supine with arms raised, and cooperate with breathholding instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with lung cancer who will undergo SBRT at USC hospitals and clinics.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Change in blood flow (mL/min/100 g) as measured on perfusion CT | Baseline to up to 3 months post SBRT
  Descriptive statistics including mean and standard deviation or median and range, will be used to summarize the distribution of perfusion parameters (blood flow, blood volume, mean transit time and permeability), as well as their changes from baseline to the time-points after SBRT. Precision of the estimated means will be provided. Line graphs will be used to display the changes in the parameters over time. If the distribution of the data permits, mixed-effect linear regression analysis will be performed to examine the patterns of the pre- vs. post-SBRT change in the endpoints.
Change in blood volume (mL/100 g) as measured on perfusion CT | Baseline to up to 3 months post SBRT
  Descriptive statistics including mean and standard deviation or median and range, will be used to summarize the distribution of perfusion parameters (blood flow, blood volume, mean transit time and permeability), as well as their changes from baseline to the time-points after SBRT. Precision of the estimated means will be provided. Line graphs will be used to display the changes in the parameters over time. If the distribution of the data permits, mixed-effect linear regression analysis will be performed to examine the patterns of the pre- vs. post-SBRT change in the endpoints.
Change in mean transit time (seconds) as measured on perfusion CT | Baseline to up to 3 months post SBRT
  Descriptive statistics including mean and standard deviation or median and range, will be used to summarize the distribution of perfusion parameters (blood flow, blood volume, mean transit time and permeability), as well as their changes from baseline to the time-points after SBRT. Precision of the estimated means will be provided. Line graphs will be used to display the changes in the parameters over time. If the distribution of the data permits, mixed-effect linear regression analysis will be performed to examine the patterns of the pre- vs. post-SBRT change in the endpoints.
Change in permeability (mL/min/100 g) as measured on perfusion CT | Baseline to up to 3 months post SBRT
  Descriptive statistics including mean and standard deviation or median and range, will be used to summarize the distribution of perfusion parameters (blood flow, blood volume, mean transit time and permeability), as well as their changes from baseline to the time-points after SBRT. Precision of the estimated means will be provided. Line graphs will be used to display the changes in the parameters over time. If the distribution of the data permits, mixed-effect linear regression analysis will be performed to examine the patterns of the pre- vs. post-SBRT change in the endpoints.

SECONDARY OUTCOMES:
Clinical tumor response assessed by CT scans as determined by Response Evaluation Criteria in Solid Tumors criteria version 1.1 | Up to 24 months post SBRT
  Descriptive statistics will also be used in the analyses of the secondary endpoints. Correlations between the endpoints will be examined with scatter plots and/or box plots. Patient's response status will be correlated with tumor perfusion parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lee, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States